CLINICAL TRIAL: NCT05011006
Title: Correlation of Circulating NT-3 Levels and Function in Individuals With Peripheral Neuropathy or Charcot-Marie-Tooth Neuropathy
Brief Title: NT-3 Levels and Function in Individuals With CMT
Status: Not yet recruiting | Type: Observational
Sponsor: Zarife Sahenk (Other)
Responsible Party: Sponsor-Investigator, Zarife Sahenk, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: 19-0353
Record Dates: First submitted 2020-03-04; First posted 2021-08-18 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Charcot-Marie-Tooth Disease; Peripheral Neuropathy; Chronic Inflammatory Demyelinating Polyneuropathy
Keywords: NT-3; CMT1A; Neuropathy
MeSH Terms: conditions — Charcot-Marie-Tooth Disease; Peripheral Nervous System Diseases; Polyradiculoneuropathy, Chronic Inflammatory Demyelinating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: NT3 blood draw — blood draw

SUMMARY:
This study will assess the serum NT-3 levels in individuals with the diagnosis of peripheral neuropathy or any type of Charcot-Marie-Tooth Neuropathy (CMT) and correlate this with function.

DETAILED DESCRIPTION:
This study will assess the serum NT-3 levels in those with a peripheral neuropathy diagnosis which will help to determine the therapeutic levels of NT-3 in subjects that will receive AAV1.NT-3 gene therapy in a future study. This study also aims to define the natural history of any type of Charcot-Marie Tooth Disease (CMT), better define the rate of disease progression and skeletal muscle involvement. Another aim is to generate a registry of well-characterized CMT patients who may be candidates for future trials.

ELIGIBILITY:
Inclusion Criteria:

* Males or females from 7 years of age or older
* Diagnosis of acquired peripheral neuropathy (PN) such as due to diabetes, chemo-induced, autoimmune chronic inflammatory demyelinating polyneuropathy (CIDP) established by a report of electrical studies or with a known genetic CMT diagnosis. Definitive diagnosis of PN is established with a report of electrical studies, EMG/nerve conduction studies.2
* Perform assessments to the best of their ability with reliable results as deemed by the evaluator.
* Ability to attend scheduled appointments
* Ability to provide informed consent (or assent for ages 9-18)

Exclusion Criteria:

* Current pregnancy per medical history
* Has a medical condition or extenuating circumstances that, in the opinion of the investigator, might compromise the subject's wellbeing, safety, or clinical interpretability

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and female subjects, from 7 years of age and over with a definitive diagnosis of acquired peripheral neuropathy or genetically determined CMT neuropathy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2027-11-13 (Estimated); Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Assess change in Manual Muscle Testing (MMT) | Compare baseline to Year 1 and Year 2 visits.
  Weakness in the major motor groups can be documented by using manual muscle testing. This exam allows the symmetry of strength, along with distribution and degree of weakness to be assessed. The Medical Research Council lists the major motor groups as: neck flexion, hip extension, knee flexion, ankle plantar flexion, and hip abduction. Depending on the clinical circumstances, the exam can be individualized. The Medical Research Council provides a scale ranging from 0-5. Inter-rater reliability will be documented by all evaluators of the trial. A rating of 5 indicates full range of motion, whereas a rating of 0 indicates no movement.
Assess change in 100 Meter Timed Test (100m): | Compare baseline to Year 1 and Year 2 visits.
  Directions for study procedures will be provided in a way the subject can understand (i.e. verbal and/or written instruction, demonstration, practice, etc.). Once the subject is comfortable with study procedures, they will complete the 100m test one time. Patients will be asked to run a set course of 25 meters for 4 laps for a total distance of 100 meters. The time to complete in seconds will be recorded.
Assess change in Timed Functional Testing: | Compare baseline to Year 1 and Year 2 visits.
  Timed Functional Testing can include time to ascend/descend 4 standard-sized stairs, time to rise from the floor (from NSAD), and the 10-meter run (from the NSAD).
Assess change in PROMIS Upper Extremity Function and Mobility Scales: | Compare baseline to Year 1 and Year 2 visits.
  The PROMIS Upper Extremity Function and Mobility instruments are patient-reported outcomes (PRO) that utilize a patient reported and/or parent proxy scale based on the patient's age that measures an individual's perceived upper extremity function and mobility.
Assess change in Abilities Captured Through Interactive Video Evaluation (ACTIVE) | Compare baseline to Year 1 and Year 2 visits.
  ACTIVE is a video game that utilizes the Microsoft Kinect camera to measure functional reaching volume while the patient is motivated to squish spiders or collect gems.
Assess change in CMT Pediatric Scale (CMTPedS) | Compare baseline to Year 1 and Year 2 visits.
  The CMTPedS is a clinician-administered scale that rates patient performance on various functional activities involving the upper extremities, lower extremities, balance, and gait. The CMTPedS generates a linear score of disability ranging from 0 (not affected) to 44 (severely affected).
Assess change in Timed Up and Go | Compare baseline to Year 1 and Year 2 visits.
  The Timed Up and Go test (TUG) is a simple test used to assess a person's mobility and requires both static and dynamic balance. It uses the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down.
Assess change in Forced Vital Capacity | Compare baseline to Year 1 and Year 2 visits.
  Forced expiratory volume (FEV) measures how much air a person can exhale during a forced breath. Forced vital capacity (FVC) is the total amount of air exhaled during the FEV test.
Assess change in Exploratory Gait Evaluation | Compare baseline to Year 1 and Year 2 visits.
  We may attempt to quantify gait using vibration sensors, activity monitors, or a portable walkway providing temporal spatial gait analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Zarife Sahenk, MD., PhD., Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No